CLINICAL TRIAL: NCT01127022
Title: Effect of Maternal Choline Intake on Maternal/Fetal Biomarkers of Choline Status
Brief Title: Effect of Maternal Choline Intake on Choline Status and Health Biomarkers During Pregnancy and Lactation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: American Egg Board (Other); National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry); USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: OSP No: 59370, 57100, 58222
Record Dates: First submitted 2010-05-17; First posted 2010-05-20 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Pregnancy; Lactation
Keywords: Pregnancy; Lactation; Choline; Cognition; Biomarkers
MeSH Terms: conditions — Breast Feeding | interventions — Choline

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 480 mg/d choline intake (Active Comparator): 480 mg/d choline derived from the diet [380 mg choline/d] plus supplemental choline chloride [100 mg choline/d]
  Interventions: Dietary Supplement: choline chloride
- 930 mg/d choline intake (Experimental): 930 mg/d choline derived from the diet [380 mg choline/d] plus supplemental choline chloride [550 mg choline/d]
  Interventions: Dietary Supplement: Choline Chloride

INTERVENTIONS:
Dietary Supplement: choline chloride — Women will consume a diet providing 380 mg/d total choline plus 100 mg/d supplemental choline [from choline chloride] for a total choline intake of 480 mg/d. The choline chloride will be administered in cran-grape juice.
  Arms: 480 mg/d choline intake
Dietary Supplement: Choline Chloride — Women will consume a diet providing 380 mg/d total choline plus 550 mg/d supplemental choline [from choline chloride] for a total choline intake of 930 mg/d. The choline chloride will be administered in cran-grape juice.
  Arms: 930 mg/d choline intake

SUMMARY:
The purpose of this study is to investigate the effect of varied maternal choline intake on maternal/fetal biomarkers of choline status, genomic expression and metabolomic profiling.

DETAILED DESCRIPTION:
Choline is a micronutrient used for the structural integrity of cell membranes, lipid transport/metabolism, methylation reactions and cholinergic neurotransmission. Prenatal and early postnatal choline exposure plays a critical role in brain development and cognition based on animal data. Although it is recognized that choline use is particularly high during pregnancy and lactation, the level of choline intake needed to optimize maternal and fetal health outcomes is unknown. The primary objective of this study was to investigate the metabolic and genomic effects of two doses of choline intake, 450 mg/d (the adequate intake level for pregnant women) and 900 mg/d in pregnant, lactating, and nonpregnant control women. A secondary objective was to examine the effect of extra maternal choline intake on the child's cognitive performance (i.e, learning, memory and attention). To accomplish these objectives, pregnant women (wk 27 gestation), nonpregnant control women, and lactating women consumed controlled choline intakes of 480 or 930 mg/d for 10 to 12 weeks. The basal diet provided 380 mg/d; supplemental choline chloride, 100 or 550 mg/d, was used to achieve the target intake levels. During the last half of the study, a small portion (~ 20%) of the total choline intake was derived from deuterium labeled choline, a stable isotope. Blood, urine and/or breast milk were collected at baseline and at select timepoints throughout the study duration. For pregnant women, a maternal blood sample was obtained at the time of delivery along with a cord blood sample and the placental tissue. Genomic and metabolomic profiling were performed on the collected biological samples along with specific measurements of choline status. Non-invasive tests assessing cognitive function were performed on the children of the pregnant and lactating study participants. This controlled feeding study has also been extended to investigate dose-response relationships for other micronutrients including folate, vitamin B12, vitamin D, and biotin.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant (wk 27 gestation) or lactating (postnatal day 30) or nonpregnant
* Healthy
* Non-smoker

Exclusion Criteria:

* Liver or kidney problems
* Alcohol or illegal drug misuse/abuse

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Maternal biomarkers of choline status | 10-12 Weeks

SECONDARY OUTCOMES:
Genomic expression as function of maternal choline intake | 10-12 Weeks
Cognitive performance in children of study participants | 12 months
Metabolomic profiling as a function of maternal choline intake | 10-12 Weeks
Biomarkers for additional micronutrients | 10-12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marie A Caudill, PhD, RD, Principal Investigator — Cornell University
Locations (1):
- Human Metabolic Research Unit, Cornell University, Ithaca, New York, United States

REFERENCES:
- [Result] Yan J, Jiang X, West AA, Perry CA, Malysheva OV, Devapatla S, Pressman E, Vermeylen F, Stabler SP, Allen RH, Caudill MA. Maternal choline intake modulates maternal and fetal biomarkers of choline metabolism in humans. Am J Clin Nutr. 2012 May;95(5):1060-71. doi: 10.3945/ajcn.111.022772. Epub 2012 Mar 14. PMID 22418088
- [Result] Jiang X, Bar HY, Yan J, West AA, Perry CA, Malysheva OV, Devapatla S, Pressman E, Vermeylen FM, Wells MT, Caudill MA. Pregnancy induces transcriptional activation of the peripheral innate immune system and increases oxidative DNA damage among healthy third trimester pregnant women. PLoS One. 2012;7(11):e46736. doi: 10.1371/journal.pone.0046736. Epub 2012 Nov 2. PMID 23133592
- [Result] Jiang X, Yan J, West AA, Perry CA, Malysheva OV, Devapatla S, Pressman E, Vermeylen F, Caudill MA. Maternal choline intake alters the epigenetic state of fetal cortisol-regulating genes in humans. FASEB J. 2012 Aug;26(8):3563-74. doi: 10.1096/fj.12-207894. Epub 2012 May 1. PMID 22549509
- [Result] West AA, Yan J, Perry CA, Jiang X, Malysheva OV, Caudill MA. Folate-status response to a controlled folate intake in nonpregnant, pregnant, and lactating women. Am J Clin Nutr. 2012 Oct;96(4):789-800. doi: 10.3945/ajcn.112.037523. Epub 2012 Aug 29. PMID 22932279
- [Result] Jiang X, Bar HY, Yan J, Jones S, Brannon PM, West AA, Perry CA, Ganti A, Pressman E, Devapatla S, Vermeylen F, Wells MT, Caudill MA. A higher maternal choline intake among third-trimester pregnant women lowers placental and circulating concentrations of the antiangiogenic factor fms-like tyrosine kinase-1 (sFLT1). FASEB J. 2013 Mar;27(3):1245-53. doi: 10.1096/fj.12-221648. Epub 2012 Nov 29. PMID 23195033
- [Result] West AA, Yan J, Jiang X, Perry CA, Innis SM, Caudill MA. Choline intake influences phosphatidylcholine DHA enrichment in nonpregnant women but not in pregnant women in the third trimester. Am J Clin Nutr. 2013 Apr;97(4):718-27. doi: 10.3945/ajcn.112.050211. Epub 2013 Feb 27. PMID 23446897
- [Derived] Bahnfleth CL, Strupp BJ, Caudill MA, Canfield RL. Prenatal choline supplementation improves child sustained attention: A 7-year follow-up of a randomized controlled feeding trial. FASEB J. 2022 Jan;36(1):e22054. doi: 10.1096/fj.202101217R. PMID 34962672
- [Derived] Klatt KC, McDougall MQ, Malysheva OV, Brenna JT, Roberson MS, Caudill MA. Reproductive state and choline intake influence enrichment of plasma lysophosphatidylcholine-DHA: a post hoc analysis of a controlled feeding trial. Br J Nutr. 2019 Dec 14;122(11):1221-1229. doi: 10.1017/S0007114519002009. PMID 31782377
- [Derived] Park H, Brannon PM, West AA, Yan J, Jiang X, Perry CA, Malysheva OV, Mehta S, Caudill MA. Vitamin D Metabolism Varies among Women in Different Reproductive States Consuming the Same Intakes of Vitamin D and Related Nutrients. J Nutr. 2016 Aug;146(8):1537-45. doi: 10.3945/jn.116.229971. Epub 2016 Jun 22. PMID 27335139
- [Derived] Davenport C, Yan J, Taesuwan S, Shields K, West AA, Jiang X, Perry CA, Malysheva OV, Stabler SP, Allen RH, Caudill MA. Choline intakes exceeding recommendations during human lactation improve breast milk choline content by increasing PEMT pathway metabolites. J Nutr Biochem. 2015 Sep;26(9):903-11. doi: 10.1016/j.jnutbio.2015.03.004. Epub 2015 Apr 15. PMID 26025328
- [Derived] Bae S, West AA, Yan J, Jiang X, Perry CA, Malysheva O, Stabler SP, Allen RH, Caudill MA. Vitamin B-12 Status Differs among Pregnant, Lactating, and Control Women with Equivalent Nutrient Intakes. J Nutr. 2015 Jul;145(7):1507-14. doi: 10.3945/jn.115.210757. Epub 2015 May 20. PMID 25995278
- [Derived] Perry CA, West AA, Gayle A, Lucas LK, Yan J, Jiang X, Malysheva O, Caudill MA. Pregnancy and lactation alter biomarkers of biotin metabolism in women consuming a controlled diet. J Nutr. 2014 Dec;144(12):1977-84. doi: 10.3945/jn.114.194472. Epub 2014 Aug 13. PMID 25122647
- [Derived] Yan J, Jiang X, West AA, Perry CA, Malysheva OV, Brenna JT, Stabler SP, Allen RH, Gregory JF 3rd, Caudill MA. Pregnancy alters choline dynamics: results of a randomized trial using stable isotope methodology in pregnant and nonpregnant women. Am J Clin Nutr. 2013 Dec;98(6):1459-67. doi: 10.3945/ajcn.113.066092. Epub 2013 Oct 16. PMID 24132975